CLINICAL TRIAL: NCT02411552
Title: Systematic Initiative to Increase Activity in Schools
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Department of Public Instruction (Unknown)
Responsible Party: Sponsor
Other Study IDs: Wisconsin Active Schools
Record Dates: First submitted 2015-03-31; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Cardiovascular Fitness
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention schools: These schools were promoting 4 strategies to increase physical activity in students.
  Interventions: Behavioral: physical activity
- Control schools: These schools continued with standard programming for activity during year 1, and implemented intervention during years 2 and 3.
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity — 4 strategies are: (1) increased activity time during physical education class, (2) active recess, (3) opportunities for activity before and after school, and (4) active classroom breaks

SUMMARY:
This initiative is a prospective study evaluating the effects of implementing physical activity strategies in Wisconsin schools with low socioeconomic status on childhood fitness.

DETAILED DESCRIPTION:
This initiative is a prospective study evaluating the effects of implementing physical activity strategies in Wisconsin schools with low socioeconomic status on childhood fitness. Forty-nine schools participated in the study providing de-identified fitness data for students for 3 consecutive years. Twenty-five schools initiated physical activity interventions in year one and 24 schools initiating physical activity interventions in year two.

ELIGIBILITY:
Inclusion Criteria:

* all children between 3rd and 8th grade

Exclusion Criteria:

* children who could not perform PACER (exercise)

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Wisconsin schools with low socio-economic status (grades 3-8)
Sampling Method: Probability Sample
Enrollment: 4894 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
PACER fitness test | performed every 6 months each school year for 3 years
  PACER is a 20 meter shuttle run in PE class

CONTACTS AND LOCATIONS:
Overall Officials: Aaron L Carrel, Principal Investigator — University of Wisconsin, Madison